CLINICAL TRIAL: NCT07047573
Title: Clinical Application Research on Differentiating Benign and Malignant Pulmonary Nodules Based on Multi-omics Detection Technology
Brief Title: Multi-omics Detection Techniques for Differentiating Benign and Malignant Pulmonary Nodules
Status: Recruiting | Type: Observational
Sponsor: Zhao Jun (Other)
Responsible Party: Sponsor-Investigator, Zhao Jun, Thoracic Surgery, The First Affiliated Hospital of Soochow University
Organization: The First Affiliated Hospital of Soochow University (Other)
Other Study IDs: 2024735
Record Dates: First submitted 2025-06-24; First posted 2025-07-02 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Lung Cancer (Diagnosis); Pulmonary Nodule Persistent
Keywords: Cancer immunotherapy; Peripheral Blood; Tumor antigen specific T cells
MeSH Terms: conditions — Lung Neoplasms; Disease | interventions — Antigens, Neoplasm

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Biological: PBMCS were isolated from the peripheral blood of hospitalized patients with pulmonary nodules and incubated with nanoparticles loaded with tumor antigens for a specific period of time to detect cancer — Research on the in vitro Stimulation of Pbmc by Tumor Antigen Nanoparticles PBMCS were isolated from the peripheral blood of hospitalized patients with pulmonary nodules and incubated with nanoparticles loaded with tumor antigens for a specific period of time to detect cancer-related T cells or cytokines in vitro. The content of this type of T cells or cytokines is positively correlated with tumors. On the contrary, the content of T cells or cytokines in patients with benign pulmonary nodules is negatively correlated with the tumor. Furthermore, the benign and malignant nature of pulmonary nodules in patients is determined through the combination of patient imaging data and clinicopathological data.

SUMMARY:
Research objective: To explore the clinical application effect of multi-omics detection based on flow cytometry analysis, single-cell data and images combined with clinical features in differentiating the benign and malignant nature of pulmonary nodules and the early diagnosis of lung cancer

DETAILED DESCRIPTION:
Research design: It is planned to collect pulmonary nodules confirmed by preoperative CT during the period from January 2021 to June 2020 The peripheral blood and clinical information of 100 patients who underwent surgical operations were classified according to the pathological diagnosis of the patients It is the malignant pulmonary nodule group and the benign pulmonary nodule group. Through single-cell sequencing, flow cytometry analysis and radiomics The purpose of identifying the benign and malignant nature of pulmonary nodules is: ① To predict the benign and malignant nature of pulmonary nodules before surgery; ② Explore evil the differences in the immune microenvironment between patients with sexual and benign pulmonary nodules, and the search for specific markers with clinical value Object ③ Compare the diagnostic sensitivity of the new prediction method with that of traditional tumor markers and explore its role as a predictor The potential for measuring the benign and malignant nature of pulmonary nodules

ELIGIBILITY:
Inclusion Criteria:

* Patient underwent a ct examination
* Patient was confirmed to have pulmonary nodules
* Patient has been determined to undergo surgical treatment
* There are clear pathological results
* The clinicopathological data are complete

Exclusion Criteria:

* Patient has no ct examination results
* Refuse surgical treatment
* Patient has no clear pathological diagnosis
* Patients with hematogenic infectious diseases, such as HIV, hepatitis B or hepatitis C.
* Patients with tumor emergencies that require immediate treatment.
* Poor vascular conditions.
* Abnormal coagulation function or receiving anticoagulant or thrombolytic therapy.
* Patients with hematogenic infectious diseases, such as HBV.
* Patients with psychiatric disorders or severe mental illnesses.
* Patients who have difficulty communicating or are unable to be followed up for a long time

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The patient must be an inpatient of our hospital, have undergone ct examination and been confirmed as having pulmonary nodules, and have received surgical treatment with a clear pathological diagnosis. The medical records are complete and available for follow-up visits.
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Changes in peripheral blood immune indicators, differences in radiomics and clinicopathological characteristics | Before surgery for patients with pulmonary nodules
Tumor antigen-specific T cells were detected by flow cytometry or single-cell sequencing to determine the differences in the immune microenvironment between patients with benign pulmonary nodules and those with malignant pulmonary nodules. | Before surgery for patients with pulmonary nodules
  Tumor antigen-specific T cells were detected by flow cytometry or single-cell sequencing to determine the differences in the immune microenvironment between patients with benign pulmonary nodules and those with malignant pulmonary nodules. The flow cytometry antibodies used to label activated T cells in this study include CD19, CD3, CD4, CD8.
  CD25, CD39, CD137,Foxp3, IFN γ, etc.

CONTACTS AND LOCATIONS:
Locations (1):
- Soochow university, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided